CLINICAL TRIAL: NCT01649102
Title: Impact of Catheter Design on Catheter Survival in Chronic Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Prof. Dr. An De Vriese, M.D., Ph. D., AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B04920108373
Record Dates: First submitted 2012-07-18; First posted 2012-07-25 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Hemodialysis; Catheter Related Bloodstream Infection; Mechanical Catheter Dysfunction
Keywords: Chronic hemodialysis; Tunneled cuffed catheter; Catheter-related bloodstream infection; Mechanical catheter dysfunction; impact of catheter design on outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palindroom catheter (Experimental): Insertion of Palindroom catheter
  Interventions: Device: Tunneled Cuffed Catheter (Palindroom, Hemoglide Bard)
- Hemoglide Bard Catheter (Experimental): Insertion of Hemoglide Bard Catheter
  Interventions: Device: Tunneled Cuffed Catheter (Palindroom, Hemoglide Bard)

INTERVENTIONS:
Device: Tunneled Cuffed Catheter (Palindroom, Hemoglide Bard) — A tunneled cuffed catheter is inserted, randomization between:
  * Palindroom
  * Hemoglide Bard

SUMMARY:
The trial aims to compare the performance of two tunneled cuffed catheters (TCC) in chronic hemodialysis patients. The design of the catheter may affect the propensity for thrombosis and hence intraluminal infection, as well the percentage of recirculation and hence the efficiency of dialysis.

DETAILED DESCRIPTION:
The use of tunneled cuffed catheters (TCCs) as vascular access is discouraged in the NKF DOQI guidelines, because of their propensity for infection, thrombosis, inadequate and/or irregular blood flow rates and damage to large central veins. In addition, emerging data suggest a link between catheter use and cardiovascular morbidity and mortality. Nevertheless, they are still frequently used in the hemodialysis population, either because of documented inadequate vascular access anatomy, or as a bridge to a functional permanent access.

A large number of TCC are available, that mainly differ with respect to material type, lumen diameter and design, tip design, as well as presence and design of side holes. There is currently no proven advantage of one long-term catheter design over another.

The design of the catheter tip may affect the propensity for thrombosis and hence intraluminal infection, as well the percentage of recirculation, especially when arterial and venous blood tubing are reversed. Commonly used catheters have a staggered tip design, meaning that the outflow tip extends several centimetres (typically a minimum of 2.5 cm) beyond the inflow tip, to prevent recirculation. Other designs are a split tip, or a symmetrical tip. In the latter type, used in the Palindrome® (Covidien) catheter, a spiral separator is incorporated allowing either lumen to be used as the arterial port.

Many catheters have multiple side holes, to decrease shear rate and increase flow on the arterial side and reflecting the belief that backup inflow is necessary in the case of obstruction. However, side holes can also promote thrombosis and infection due to the irregularity of their cut surfaces. Especially the distal side holes comprise a low flow zone with an increased clotting risk. The Palindrome® (Covidien) catheter has laser cut side holes, which are thought to have a smoother surface and a lower tendency to cause thrombosis.

Inadequate blood flow in a catheter is often mended by reversal of the inlet and outlet lumens. However, reversal of flow leads to a substantial increase of recirculation (from 2%-3% to 10%), affecting the efficiency of treatment. It should therefore never be used except temporarily until the problem is definitively corrected. The symmetrical tip design of the Palindrome® (Covidien) catheter allows lumen reversal without increased recirculation.

The present randomized controlled trial (RCT) is designed to evaluate in chronic hemodialysis patients the performance of two TCC with different design: the Palindrome® (Covidien), which is a symmetrical spiral z-tip catheter made from carbothane and the Hemoglide® (Bard), which has a 3 cm staggered tip and is made of polyurethane.

ELIGIBILITY:
Inclusion Criteria:

All patients (male or female, age < 18 years) on chronic hemodialysis who require a tunneled cuffed catheter as temporary or definite vascular access are eligible. Written informed consent is required prior to inclusion.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Life-expectance of < 6 months due to major co-morbid conditions
* Inability to provide informed consent
* Occlusion or inaccessibility of the right internal jugular vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
overall catheter survival rate | 3 years

SECONDARY OUTCOMES:
Mechanical catheter dysfunction: number of dialysis sessions requiring urokinase administration per 1000 catheter days; number of catheter removals for mechanical obstruction | 3 years

OTHER OUTCOMES:
Dialysis efficiency: Kt/V; mean achieved blood flow rate per dialysis session | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: An S De Vriese, M.D., Ph.D., Principal Investigator — AZ ST JAN Brugge Oostende AV
Locations (1):
- AZ ST JAn Brugge Oostende AV, Bruges, Belgium